CLINICAL TRIAL: NCT06865157
Title: Bolsillo Saludable: Feasibility of a Healthy Food Subsidy on Healthy Eating in Low-Income Households in Chile
Brief Title: Healthy Food Subsidy Project in Chile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Bloomberg Philanthropies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5128637; 5128637 (Other Grant/Funding Number: Bloomberg Philanthropies)
Record Dates: First submitted 2024-11-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: Feasibility Studies; Food Security
Keywords: Chile; Fruit and vegetables subsidy; Feasibility study

STUDY DESIGN:
Intervention Model Description: The Healthy Wallet program is a mobile-based initiative designed to promote healthy eating among low-income families by incentivizing the purchase of fruits and vegetables at open markets. Over the course of two months, 30 families received monthly benefits redeemable at participating stalls within the Juan Pinto Durán open market in Santiago, Chile. Registered vendors prominently displayed a distinctive Healthy Wallet identification sign with a unique code, ensuring easy identification. Beneficiaries used the mobile app to check their available funds and complete purchases by entering the stall code. Meanwhile, vendors utilized their own app to track sales and maintain transaction records, streamlining the invoicing process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy Wallet (Experimental): Each eligible household receives a monthly electronic transfer of 16,000 CLP (approximately USD 17) per eligible member to purchase fruits and vegetables from authorized vendors at the Juan Pinto Durán open market. A dedicated mobile application manages the process by crediting the benefit to participants' accounts, simplifying its use at the market, and ensuring seamless payment to vendors.
  Interventions: Other: Healthy Wallet

INTERVENTIONS:
Other: Healthy Wallet — The Healthy Wallet program is a mobile-based initiative designed to promote healthy eating among low-income families by incentivizing the purchase of fruits and vegetables at open markets. Over a two-month period, 30 families received monthly benefits to use at a designated open market.

SUMMARY:
Feasibility Study

Objective:

The objective of this feasibility study is to develop and evaluate the feasibility and acceptability of a healthy food subsidy program within the Chilean context. The program, called Healthy Wallet, is a smartphone app-based initiative aimed at incentivizing low-income families to purchase fruits and vegetables at open markets. The findings from this study are intended to inform and potentially accelerate the implementation of similar policies in other countries.

Methods:

This study assessed the feasibility of implementing the Healthy Wallet subsidy program, designed to promote healthy eating habits among low-income families. The program incentivized the purchase of fruits and vegetables at local ferias (open markets) and was delivered through a smartphone application. The research adopted a community-based approach, leveraging existing social support systems to identify eligible beneficiaries and streamline the distribution of benefits. Open markets served as redemption sites for the subsidies.

The study engaged 30 families and 8 vendors in an 8-week pilot program conducted from June to August 2024. Data collection included pre- and post-implementation surveys, as well as focus group discussions: three with participating families and one with vendors. These methods aimed to evaluate the app's effectiveness, user experience, and overall feasibility of the program. Insights from the study will guide recommendations for scaling the initiative to a national level and beyond.

DETAILED DESCRIPTION:
Study Design:

This study employed an eight-week feasibility approach (Healthy Wallet) utilizing a mixed-methods assessment. The quantitative component consisted of a pre-post single-arm study, while the qualitative component involved focus group discussions with both vendors and participants.

Intervention:

The Healthy Wallet program is a mobile-based initiative aimed at promoting healthy eating habits among low-income families by incentivizing the purchase of fruits and vegetables at open markets. The program provides a monthly electronic transfer of 16,000 CLP (approximately 17 USD) for each eligible household member, including children under 18, students under 25, and individuals with disabilities. The primary food purchaser in each household receives the transfer, which is exclusively redeemable at registered stalls in the open market.

To ensure seamless transactions, registered vendors display a distinctive Healthy Wallet identification sign with a unique code. Beneficiaries use the mobile application to view available funds and complete purchases by entering the vendor's stall code. A separate vendor application tracks sales and maintains transaction records for efficient invoicing.

Sample:

The program engaged 30 families, who received monthly benefits for two consecutive months to use at 6 participating stalls within the Juan Pinto Durán open market.

Eligibility Criteria:

Eligibility aligned with Chile's existing social protection framework, leveraging the Emergency Family Wallet government subsidy established to address rising food prices during the COVID-19 pandemic. Households that participated in the Emergency Family Wallet program (2023-2024) were eligible.

The designated household representative, responsible for receiving and managing the benefit, had to meet the following criteria:

Be at least 18 years old (legal age). Be a parent or guardian of a child aged 0-5 years. Be responsible for household grocery purchases. Vendors operating at the Juan Pinto Durán open market were excluded from household eligibility.

Subsidy Delivery Platform:

A private mobile application, originally developed for university food benefits, was adapted for this pilot program. A private company managed the entire process, including loading benefits into participants' accounts, facilitating their use at the Juan Pinto Durán open market, and ensuring payment to vendors. This company provided its services pro bono, offering technical expertise and logistical support at no cost.

Ethical Considerations:

The study was conducted in accordance with the Declaration of Helsinki. The protocol and informed consent forms were approved by the Ethics Committee of the Faculty of Medicine, University of Chile.

ELIGIBILITY:
Inclusion Criteria:

Households that are beneficiaries of the Bolsillo Familiar Electrónico program in 2023-2024 and have children under 5 years of age.

Availability to shop at the local open-air market (feria libre).

Exclusion Criteria:

Individuals who are market vendors (feria vendors).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of the monetary subsidy spent daily by each household, based on the records from the subsidy delivery platform. | Daily throughout the two months of follow-up
  Percentage of the monetary subsidy spent daily by each household, based on the records from the subsidy delivery platform.
Percentage of households that used the monetary subsidy at least once per month, based on the records from the subsidy delivery platform | Weekly throughout the two months of follow-up
  Percentage of households that used the monetary subsidy at least once per month, based on the records from the subsidy delivery platform
Perceived utility of the subsidy program among beneficiaries, evaluated through online surveys | At the end of the study, at two months of follow-up
  Perceived utility of the subsidy program among beneficiaries, evaluated through online surveys (Likert scale)
Perceived utility of the subsidy program among vendors, evaluated through online surveys | At the end of the study, at two months of follow-up
  Perceived utility of the subsidy program among vendors, evaluated through online surveys (Yes/No questionnaire)
Self-reported satisfaction of the subsidy program among beneficiaries, evaluated through focus groups | At the end of the study, at two months of follow-up
  Self-reported satisfaction of the subsidy program among beneficiaries, evaluated through focus groups
Self-reported satisfaction of the subsidy program among vendors, evaluated through focus groups | At the end of the study, at two months of follow-up
  Self-reported satisfaction of the subsidy program among vendors, evaluated through focus groups
Perceived utility of the subsidy platform among beneficiaries, evaluated through online surveys | At the end of the study, at two months of follow-up
  Perceived utility of the subsidy program among beneficiaries, evaluated through online surveys (Likert scale)
Perceived utility of the subsidy platform among vendors, evaluated through online surveys | At the end of the study, at two months of follow-up
  Perceived utility of the subsidy program among vendors, evaluated through online surveys (Yes/No questionnaire)
Self-reported satisfaction of the subsidy platform among beneficiaries, evaluated through focus groups | At the end of the study, at two months of follow-up
  Self-reported satisfaction of the subsidy platform among beneficiaries, evaluated through focus groups
Self-reported satisfaction of the subsidy platform among vendors, evaluated through focus groups | At the end of the study, at two months of follow-up
  Self-reported satisfaction of the subsidy platform among vendors, evaluated through focus groups

OTHER OUTCOMES:
Self-reported monthly expenditure on all fruits purchased from the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly expenditure on all fruits purchased from the open market, based on a questionnaire
Self-reported monthly expenditure on all vegetables purchased at the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly expenditure on all vegetables purchased at the open market based on a questionnaire
Self-reported monthly expenditure on all fruits and vegetables combined, purchased from the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly expenditure on all fruits and vegetables combined, purchased from the open market, based on a questionnaire
Self-reported monthly combined fruit and vegetable purchases (in kilograms) from the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly combined fruit and vegetable purchases (in kilograms) from the open market, based on a questionnaire
Self-reported monthly fruit purchases (in kilograms) at the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly fruit purchases (in kilograms) at the open market, based on a questionnaire
Self-reported monthly vegetable purchases (in kilograms) at the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly vegetable purchases (in kilograms) at the open market, based on a questionnaire
Self-reported monthly vegetable purchases (in units) at the open market, based on a questionnaire | At baseline and at the end of the study (0 and 2 months of follow-up)
  Self-reported monthly vegetable purchases (in units) at the open market, based on a questionnaire
The Global Dietary Recommendations (GDR) score from the Diet Quality Questionnaire (DQQ), range 0-18 | At baseline and at the end of the study (0 and 2 months of follow-up)
  The Global Dietary Recommendations (GDR) score is a score with a range from 0 to 18 that indicates adherence to global dietary recommendations, which include dietary factors protective against non-communicable diseases (NCD). The higher the GDR score, the more recommendations are likely to be met. The GDR score is based on food group consumption during the past day and night. The GDR score is calculated as follows: NCD-Protect - NCD-Risk + 9 = GDR score It is expressed as the average score for the population.
The Non-Communicable Disease-protect (NCD-protect) score from the Diet Quality Questionnaire (DQQ), range 0-9 | At baseline and at the end of the study (0 and 2 months of follow-up)
  An indicator of dietary factors protective against non-communicable diseases (NCD) (articulated by the World Health Organization):
  * At least 400g of fruits and vegetables per day
  * Whole grains, pulses, and nuts or seeds
  * At least 25g of fiber per day The NCD-Protect score is a score with a range from 0 to 9. It is a sub-component of theGDR score, and reflects adherence to global dietary recommendations on healthy components of the diet. The NCD-Protect score is based on food consumption from 9 healthy food groups during the past day and night. A higher score indicates inclusion of more health-promoting foods in the diet, and correlates positively with meeting global dietary recommendations. It is expressed as the average score for the population.
The Non-Communicable Disease-risk (NCD-risk) score from the Diet Quality Questionnaire (DQQ), range 0-9 | At baseline and at the end of the study (0 and 2 months of follow-up)
  An indicator of dietary factors for Non-Communicable Diseases (NCD): Less than 10% (ideally less than 5%) of total energy from free sugars; Less than 10% of total energy from saturated fat, and less than 30% from total fat; Less than 5g of salt per day; Little if any processed meat, and red meat limited to no more than 350-500g per week. It is a score with a range from 0 to 9. It is a sub-component of the GDR score, and reflects adherence to global dietary recommendations on components of the diet to limit or avoid. A higher score indicates higher consumption of foods and drinks to avoid or limit, and correlates negatively with meeting global dietary recommendations. The NCD-Risk score is based on food consumption from 8 food groups to limit or avoid during the past day and night (one food group, processed meat, is double weighted). This is a negative indicator, and is expressed as the average score for the population.
The Food Group Diversity Score (FGDS) from the Diet Quality Questionnaire (DQQ), range 0-10 | At baseline and at the end of the study (0 and 2 months of follow-up)
  The Food group diversity score (FGDS) is a semicontinuous score ranging from 0 to 10, by summing the scores for each food group (0: not consumed; 1: consumed) using the following 10 food groups: 1) grains, white roots and tubers, and plantains; 2) pulses (beans, peas, and lentils); 3) nuts and seeds; 4) milk and milk products; 5) meat, poultry, and fish; 6) eggs; 7) dark green leafy vegetables; 8) other vitamin A-rich fruits and vegetables; 9) other vegetables; and 10) other fruits. The FGDS is a proxy indicator of micronutrient adequacy for the general population expressed as the mean population score.

CONTACTS AND LOCATIONS:
Overall Officials: Camila Corvalan, PhD, Principal Investigator — Institute of Nutrition and Food Technology, University of Chile
Locations (1):
- Feria Libre Juan Pinto Durán, Santiago, Macul, Chile

IPD SHARING:
Plan to Share IPD: Yes
All IPD data related to study protocol, statistical analysis plan and informed consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary results
Access Criteria: Access to IPD data will be available for qualified researchers for scientific purposes that meet specific criteria: ethical, security and administrative criteria

REFERENCES:
- [Background] Huangfu P, Pearson F, Abu-Hijleh FM, Wahlich C, Willis K, Awad SF, Abu-Raddad LJ, Critchley JA. Impact of price reductions, subsidies, or financial incentives on healthy food purchases and consumption: a systematic review and meta-analysis. Lancet Planet Health. 2024 Mar;8(3):e197-e212. doi: 10.1016/S2542-5196(24)00004-4. PMID 38453385
- [Background] Andreyeva T, Marple K, Moore TE, Powell LM. Evaluation of Economic and Health Outcomes Associated With Food Taxes and Subsidies: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Jun 1;5(6):e2214371. doi: 10.1001/jamanetworkopen.2022.14371. PMID 35648401
- [Background] Berkowitz SA, Curran N, Hoeffler S, Henderson R, Price A, Ng SW. Association of a Fruit and Vegetable Subsidy Program With Food Purchases by Individuals With Low Income in the US. JAMA Netw Open. 2021 Aug 2;4(8):e2120377. doi: 10.1001/jamanetworkopen.2021.20377. PMID 34379125